CLINICAL TRIAL: NCT01712529
Title: Effect of Supervised Physical Exercise on Endothelial Function and Endothelial Progenitor Cells in Patients With Systemic Lupus Erythematosus
Brief Title: Physical Exercise, Endothelial Function and Progenitor Endothelial Cells in Systemic Lupus Erythematosus Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Emilia Inoue Sato, Professor, PHD, Federal University of São Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09295-5
Record Dates: First submitted 2012-10-20; First posted 2012-10-23 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic lupus erythematosus; endothelium; exercise
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supervised physical exercise (Experimental): Walking at speed of the ventilatory threshold-1 heart rate obtained from cardiopulmonary exercise test and monitored by frequency meter.
  Interventions: Behavioral: Supervised physical exercise
- No supervised physical exercise (No Intervention): No intervention for 16 weeks

INTERVENTIONS:
Behavioral: Supervised physical exercise — Women with systemic lupus erythematosus with availability to perform physical exercise were allocated in exercise group (EG) to practice supervised physical exercise for one hour, three times a week for 16 weeks. Those who were not available for this activity were allocated in the control group (CG). Intervention consisted of walking at speed of the ventilatory threshold-1 heart rate obtained from cardiopulmonary exercise test and monitored by frequency meter.
  Arms: Supervised physical exercise

SUMMARY:
The purpose of this study is to evaluate the effect of supervised physical exercise on endothelial function and number of endothelial progenitor cells (EPCs) in patients with systemic lupus erythematosus, as well as evaluate the effect of supervised physical exercise on endothelium derived growth factor (VEGF) levels, disease activity, quality of life, fatigue, perceived exertion and cardiopulmonary exercise test variables.

DETAILED DESCRIPTION:
Several studies have shown that cardiovascular morbimortality is more frequent and early in SLE patients than in the general population and cardiovascular disease is an important cause of morbidity and mortality in systemic lupus erythematosus patients. Disturbances in endothelial function are implicated in its pathogenesis. Endothelial function also depends on endothelial progenitor cells (EPCs) that enhance angiogenesis, promote vascular repair and have potential as a marker of cardiovascular disease. Systemic lupus erythematosus patients have endothelial dysfunction and fewer EPCs. There are studies showing improvement of endothelial function and EPCs after physical exercise program in individuals with heart failure, diabetes and coronary arterial disease, but there isn't studies evaluating endothelial function and EPCs after.

ELIGIBILITY:
Inclusion Criteria:

* female systemic lupus erythematosus patients
* 18 to 45 years of age
* Fulfilled at least four criteria classification for lupus (ACR criteria, 1997) - Signed the consent form approved by the ethics committee of the institution

Exclusion Criteria:

* Hemoglobin < 10 mg/dL
* Neuropsychiatric, pulmonary, articular or vascular damage that would prevent the practice of exercise
* Coronary disease or heart failure, functional class ≥ II
* Pulmonary hypertension
* Uncontrolled hypertension
* Creatinine ≥ 1.4 mg/dL
* Body mass index (BMI) ≥ 35 kg/m2
* Diabetes mellitus
* Uncontrolled hypothyroidism
* Smoking in the last 12 months
* Pregnancy
* Menopause
* Use of statins in the last three months
* Practice of physical exercise in past three months
* Overlap with other autoimmune rheumatic diseases, except antiphospholipid syndrome.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2010-09; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Endothelial function and endothelial progenitor cells (EPCs) number | 16 weeks
  Patients were evaluated at baseline and after 16 weeks by high-resolution ultrasound of brachial artery in resting conditions, after reactive hyperaemia (flow-mediated dilation-FMD) and after oral glyceryl trinitrate to assess endothelial function; EPCs were evaluated by flow cytometry using anti-CD34 (cluster of differentiation 34) (FITC), anti-CD133 (PE) and anti-kinase domain receptor (KDR) (APC)

SECONDARY OUTCOMES:
Quality of life | 16 weeks
  Short Form-36
Vascular endothelial growth factor (VEGF) | 16 weeks
  ELISA
Disease activity | 16 weeks
  Systemic Lupus Erythematosus Disease Activity Index (SLEDAI)
perceived exertion | 16 weeks
  Borg scale
Fatigue | 16 weeks
  Severity fatigue scale
Ergospirometric variables | 16 weeks
  Cardiopulmonary exercise test

CONTACTS AND LOCATIONS:
Overall Officials: Emilia I Sato, MD, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] dos Reis-Neto ET, da Silva AE, Monteiro CM, de Camargo LM, Sato EI. Supervised physical exercise improves endothelial function in patients with systemic lupus erythematosus. Rheumatology (Oxford). 2013 Dec;52(12):2187-95. doi: 10.1093/rheumatology/ket283. Epub 2013 Aug 22. PMID 23970541